CLINICAL TRIAL: NCT06861556
Title: Pediatric Transversus Abdominis Plane Block Versus Quadratus Lumborum Block: a Prospective Randomized Study in Sub-umbilical Peripheral Surgery
Brief Title: Transversus Abdominis Plane Lock Versus Quadratus Lumborum Block in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tunis University (Other)
Responsible Party: Principal Investigator, Mehdi Trifa, Full Professor of Anesthesiology and Intensive Care, head chief of the department of Anesthesia and Intensive Care, Tunis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 222022
Record Dates: First submitted 2024-11-24; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Peripheral Nerve Block; Post Operative Analgesia; Ultrasound-guided Regional Anesthesia
Keywords: Transversus Abdominis Plane block; QUADRATUS LUMBORUM BLOCK; post operative analgesia; Ultrasound; Children

STUDY DESIGN:
Intervention Model Description: The patients were randomly assigned into two groups to receive after a standardized general anesthesia induction either an ultrasound-guided TAP block or Quadratus Lumborum block with 0.2ml/kg bupivacaine 0.25%
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP block group (Active Comparator): Ultrasound-guided TAP block group
  Interventions: Procedure: Ultrasound guided Transversus Abdominis Plane block with 0.2ml/kg bupivacaine 0.25%
- QLB block group (Active Comparator): Ultrasound-guided Quadratus Lumborum block group
  Interventions: Procedure: Ultrasound-guided Quadratus Lumborum block with 0.2ml/kg bupivacaine 0.25%

INTERVENTIONS:
Procedure: Ultrasound guided Transversus Abdominis Plane block with 0.2ml/kg bupivacaine 0.25% — The operator applied a linear ultrasound probe transversally to the mid-axillary line between the costal margin and iliac crest. Landmarks were then identified as three muscles layers beneath the subcutaneous tissue; from external to internal lay respectively the external oblique muscle (EO), the internal oblique muscle (IO) and the transversus abdominis (TA). The needle was inserted in plane from the iliac crest level on the midaxillary line advancing towards the midline to the fascia laying between the IO and the TA muscles until pop detection. A clear aspiration ruled out vascular effraction. Finally, the space between the two muscle planes was hydrodissected with the bupivacaine.The end goal was visualizing the IO moving upward leaving room to a hypoechoic lens-shaped local anesthetic distribution.
  Arms: TAP block group
Procedure: Ultrasound-guided Quadratus Lumborum block with 0.2ml/kg bupivacaine 0.25% — The patient was laid in a lateral decubitus position. The operator applied the probe transversally on the iliac crest directing the indicator to display the back muscles encompassed by the thoracolumbar fascia (TLF).The intended image was spotted by the emergence of the transverse process L4, delimiting the stem of a shamrock-like shape. Quadratus lumborum (QL) muscle represented the upper leaf of the shamrock, and psoas major (PM) and erector spinae (ES) stood respectively for the anterior and posterior leaves. The needle was inserted in plane from the postero-median lumbar wall directed antero-laterally with tip aiming at the posterior border of the QL muscle adjacent to the ES muscles. Pop detection indicated the middle TLF where the local anesthetic would spread, homogenous and resistance-free
  Arms: QLB block group

SUMMARY:
Although abdominal wall surgeries are also as routinely performed on pediatric patients, postoperative pain in children has remained under-researched compared to adults. Consequently, there has been a growing need for adapting regional analgesia to this distinct population. While the Transversus Abdominis Plane Block (TAPB) and Quadratus Lumborum Block (QLB) have been established as potent sensory blocks in adult practice, data on their efficiency in pediatric abdominal parietal surgeries remain scarce.

The investigators aimed to compare the analgesic effect of lateral TAPB versus posterior QLB in children undergoing elective abdominal wall surgery.

DETAILED DESCRIPTION:
Randomized controlled trial, including pediatric patients aged from 1 to 10 years old scheduled for an elective outpatient open sub-umbilical abdominal wall surgery.

After a standardized anesthesia induction protocol, patients were randomized into two parallel groups receiving either a lateral TAPB or a posterior QLB.

The investigators determined the time to first rescue analgesia as the primary outcome of the present trial. As for secondary outcomes, the investigators set out to comparatively assess block failure rates, intra operative hemodynamic features pain scores consisting of FLACC scale values, analgesic consumption attested by the number of administrated rescue paracetamol doses along the cumulative administered dose per kilogram of weight within the first postoperative 24 hours, as well as the incidence of side effects namely systemic local anesthetic toxicity symptoms, PONV, urinary retention, ICU admission or re-intervention for block-related complications.

ELIGIBILITY:
Inclusion Criteria:

* We included patients aged from 1 to 10 years old with American Society of Anesthesiologists (ASA) physical status I or II.

Exclusion Criteria:

* Non-inclusion criteria were a priorly known allergy to local anesthetics, a priorly known or suspected coagulopathy, inflammation or infection at the needle injection site, cognitive impairment preventing standard pain assessment and associated circumcision or scrotal incision.
* Later on after allocation, patients were excluded for block failure or major perioperative complications

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Time to first rescue analgesia | 3 hours
  Time (in minutes) from the completion of the block to first analgesia administration based on postoperative pain score (assessed using FLACC (Face Legs Activity Crying Consolability) in ward >3)

SECONDARY OUTCOMES:
block Failure rate | 30 minutes
  percentage of failed blocks in both groups
FLACC scale pain scores | 2 hours
  Post operative analgesia was assessed using the following measures:
  - pain scores including the Face, Legs, Activity, Cry, and Consolability (FLACC) scale, recorded at H0, H1, H2
PPMP scale scores | 24 hours
  Parents' Postoperative Pain Measure scores after discharge (at H6, H12, and H24 post operative).
Total analgesic consumption | 24 hours
  determined by the total number of rescue paracetamol doses administered (mg per kilogram of weight)
Post operative nausea and vomiting (PONV) | 24 hours
  incidence (percentage) of post operative nausea and vomiting in both groups
Urinary retention | 24 hours
  incidence (percentage) of post operative Urinary retention in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Bechir Hamza Children's Hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No